CLINICAL TRIAL: NCT02663323
Title: MeRes-1 Extend: A Prospective, Multinational, Multicenter, Single Arm, Open Label, Pilot Clinical Study of MeRes100 Sirolimus Eluting Bioresorbable Vascular Scaffold System in the Treatment of De-novo Native Coronary Artery Lesions
Brief Title: Pilot Clinical Study of MeRes100 Sirolimus Eluting Bioresorbable Vascular Scaffold System
Acronym: MeRes-1Extend
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MER/EX
Record Dates: First submitted 2015-12-07; First posted 2016-01-26 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; MeRes-1 Extend; MeRes100; Sirolimus Eluting Bioresorbable Vascular Scaffold System
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Single intervention with MeRes100 Device
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MeRes100 - BRS (Experimental): MeRes100 Sirolimus Eluting Bioresorbable Vascular Scaffold System
  Interventions: Device: MeRes100 Sirolimus Eluting Bioresorbable Vascular Scaffold System

INTERVENTIONS:
Device: MeRes100 Sirolimus Eluting Bioresorbable Vascular Scaffold System — MeRes100 Sirolimus Eluting Bioresorbable Vascular Scaffold System in the treatment of de-novo coronary artery lesions.

SUMMARY:
MeRes-1 Extend study is designed as prospective, multinational, multicentre, single arm, open label, pilot study to assess the safety and performance of the MeRes100 Sirolimus Eluting Bioresorbable Vascular Scaffold System (BRS) in subjects with de novo native coronary artery lesions. 64 subjects will be enrolled from the 8 centers located in Asia Pacific, Europe, Brazil and South Africa. Primary outcome of study will be Proportion of population reporting Major Adverse Cardiac Events at 6 months from the day of index Procedure.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Male or female subjects ≥ 18 years of age
2. Subject is able to sign written Informed Consent Form (ICF)
3. Subjects with symptomatic myocardial ischemia, chronic stable angina
4. The patient has planned intervention of a single de novo lesion in native epicardial vessel
5. Subject who is an acceptable candidate for Coronary Artery Bypass Grafting (CABG)
6. Subject is not participating in any other clinical investigation/study and agrees not to participate in any other clinical investigation/study for a period of 3 years following the index procedure.
7. Subject must agree to undergo all clinical investigation plan-required follow-up visits, angiograms and OCT as per protocol.

Angiographic Inclusion Criteria:

1. Subject with maximum two treatable de novo lesions located maximum one per native epicardial vessel located in major artery or branch, with reference vessel diameter between 2.75, 3.00 and 3.5 mm by on line QCA.
2. Target lesion length ≤ 20 mm.
3. Subjects with Lesion(s), with a visually estimated stenosis of ≥ 50% and < 100% with a TIMI flow of ≥ 1.

Exclusion Criteria:

General Exclusion Criteria:

1. Subjects unable to provide written informed consent.
2. Pregnant or nursing mother and those who plan pregnancy during the clinical investigation (female patients must have a negative pregnancy test done within 7 days prior to the index procedure and effective contraceptive must be used during participation in this clinical investigation).
3. Subjects with known allergy to Poly-L-Lactide (PLLA), Poly-D,L-Lactide (PDLLA), Sirolimus (Rapamycin) or its any analog or derivative, clopidogrel, ticlopidine, prasugrel, contrast media, platinum, ticagrelor and any drug in dual antiplatelet therapy including aspirin, both heparin and bivalirudin.
4. Subject diagnosed with Acute Myocardial Infarction (AMI) within 7 days preceding the index procedure, as indicated by elevated levels of cardiac enzymes and/or ST segment changes in Electro Cardio Gram (ECG).
5. Subject with history of previous revascularization procedures including CABG and Percutaneous Coronary Intervention (PCI).
6. Subject with vascular aneurysms, cardiac arrhythmias, congestive cardiac failure having LVEF < 30%, cardiac tamponade.
7. Recipient of an organ in an organ transplant procedure or is on a waiting list for any organ transplant.
8. Subjects receiving immunosuppression therapy or having known immunosuppressive or autoimmune disease.
9. Subjects with history of stroke, Cerebro Vascular Accident (CVA) or Transient Ischemic neurological Attack (TIA). Patients with renal insufficiency where creatinine levels are more than 1.3 mg/dl, known aplastic anaemia, chronic liver disease, platelet count <100,000 cells/mm3, a WBC of < 3,000 cells/mm3.
10. Subjects planned for elective surgery within the first 12 months after the procedure that will require discontinuing dual antiplatelet therapy
11. Subject has a history of bleeding diathesis or coagulatory disease, refuses blood transfusion, significant gastrointestinal or urinary bleed within the past 12 months.
12. Subject having extensive peripheral vascular disease that precludes safe 6F sheath insertion.
13. Subject having a history of paradoxical exercise induced vasoconstriction that is consistent with myocardial bridging in the coronary anatomy.
14. Subjects participating in another clinical investigation.
15. Subjects with short life expectancy such as cancer, Human Immunodeficiency Virus (HIV)/Acquired Immune Deficiency Syndrome (AIDS), or other co-morbid conditions that would limit compliance with the follow-up schedule of the study.

Angiographic Exclusion Criteria:

1. Subjects who are non-candidates for PCI.
2. Any of the target lesions meets any of the following criteria:

   1. Aorto-ostial location (within 3 mm)
   2. Lesion located in left main coronary artery
   3. Lesion located within 2 mm of origin of the LAD or LCx
   4. Lesion that involves a bifurcation with a side branch ≥ 2mm in diameter and ostial lesion > 40% stenosed by visual estimation or side branch requiring intervention
   5. Total occlusion (TIMI Flow 0), prior to wire crossing
   6. Extreme tortuosity proximal to or within the lesion
   7. Lesions having heavy calcification
   8. Extreme angulation (≥ 90 %) proximal to or within the lesion
3. Evidence of previous revascularization:

   1. Previous PCI with or without restenosis from previous intervention
   2. Arterial or venous graft with or without lesion located within the graft or distal to a diseased arterial or saphenous vein graft
4. The target vessel contains visible thrombus.
5. Another (clinically significant or potentially significant) lesion left untreated within target vessels (including side branch) or another significant vessel.
6. Subject requiring or potentially requiring interventional procedures other than pre-dilatation and study device implantation and post dilatation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2020-07-05 (Estimated)

PRIMARY OUTCOMES:
Primary Clinical Endpoint: Proportion of population reporting with Major Adverse Cardiac Event at 6 months from the day of index procedure. | 6 Month
Primary Safety Endpoint: Proportion of population reporting with Ischemia Driven Major Adverse Cardiac Event (ID MACE) reporting at 6 months (180 days) from the day of index procedure | 6 Month

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Alexandre Abizaid, Principal Investigator — Dante Pazzanese Hospital, Sao Paulo, Brazil
Locations (4):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil
- Medistra Hospital, Jakarta, Indonesia
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- University Clinic of Cardiology, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abizaid A, Kedev S, Ali RBM, Santoso T, Cequier A, van Geuns RVG, Chevalier B, Hellig F, Costa R, Onuma Y, Costa JR Jr, Serruys P, Bangalore S. Imaging and 2-year clinical outcomes of thin strut sirolimus-eluting bioresorbable vascular scaffold: The MeRes-1 extend trial. Catheter Cardiovasc Interv. 2021 Nov 15;98(6):1102-1110. doi: 10.1002/ccd.29396. Epub 2020 Dec 2. PMID 33269506